CLINICAL TRIAL: NCT03986918
Title: Survivorship and Patient Outcomes of Primary Total Hip Arthroplasty With the Ovation Hip System
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ortho Development Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: P-17-0013B
Record Dates: First submitted 2019-06-07; First posted 2019-06-14 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Joint Diseases; Osteoarthritis, Hip; Rheumatoid Arthritis; Psoriatic Arthritis; Avascular Necrosis of Hip
MeSH Terms: conditions — Joint Diseases; Osteoarthritis, Hip; Arthritis, Rheumatoid; Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Ovation and Ovation Tribute: All patients having undergone a total hip arthroplasty that received the Ovation® or Ovation Tribute® (Ortho Development, Draper, Utah) Hip system will be sent the survey.
  Interventions: Device: Routine Total Hip Arthroplasty

INTERVENTIONS:
Device: Routine Total Hip Arthroplasty — Patients undergoing routine total hip arthroplasty will receive surveys regarding survivorship and outcomes.

SUMMARY:
The objective of this study is to evaluate patient outcomes in regards to safety and effectiveness based on the clinical performance of the reference devices to further support the assessment of residual risk identified in the Clinical Evaluation Report for the Ortho Development Hip System.

DETAILED DESCRIPTION:
Long term surveillance of survivorship and complications can help to identify pre-surgical comorbidities, perhaps leading to a lower risk of implant failure and subsequent revision surgery. By understanding the role of comorbidities in the specific population, it is possible to increase patient outcomes and satisfaction, while reducing the costs associated with complications and revision surgeries.

This study consists of prospective collection and analysis of data for a consecutive series of patients that underwent total hip arthroplasty with the Ortho Development Ovation® Hip System at the study site between 2012 and December 2015. It is estimated that over 400 patients received the subject system. Each of these patients will receive a survey within the mail when they approach, or have exceeded, their five-year post-surgical time period.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years of age
* Patient is five years post total hip arthroplasty
* Patient received the Ovation® or Ovation Tribute® femoral stem with associated acetabular and femoral components
* Patient agrees to participate in the survey.

Exclusion Criteria:

* Patient does not have the Ovation® or Ovation Tribute® femoral stem with associated acetabular and femoral components

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Identification will occur from a list of patients having undergone total hip arthroplasty at Straub Medical Center between 2012 and the end of December 2015. Identified patients will then be screened for eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Survivorship - The number of revision surgeries over time. | 5 - 10-year follow-up
  The primary outcome will be 5-10 year survivorship of implant components, with failure defined as revision of any component.

SECONDARY OUTCOMES:
Pain and Function | 5 - 10 year follow-up
  The Hip Disability and Osteoarthritis Outcome score - joint replacement (HOOS JR) will be used. The HOOS-JR is a joint replacement survey designed to measure pain and function.
General Health | 5 - 10 year follow-up
  The Veterans Rand - 12 (VR-12) will be used to measure general health, including the ability to carry out usual activities.
Patient satisfaction. | 5 - 10 year follow-up
  A four question patient satisfaction survey will be used to measure the patient's satisfaction with their surgery, pain control, function, and ability to participate in recreational activities.

CONTACTS AND LOCATIONS:
Overall Officials: Cass Nakasone, MD, Principal Investigator — Hawai'i Pacific Health
Locations (1):
- Straub Medical Center, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No